CLINICAL TRIAL: NCT03165838
Title: Effectiveness of Shortened Time Interval to Postpartum Visit in Improving Postpartum Attendance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HM20000032
Record Dates: First submitted 2017-05-08; First posted 2017-05-24 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Pregnancy Related; Contraception; Contraception Behavior; Contraception Use
Keywords: postpartum; pregnancy; contraception; RROP
MeSH Terms: conditions — Contraception Behavior | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postpartum Visit 3-4 Weeks (Experimental): Participants will have postpartum visit scheduled 3-4 weeks after birth
  Interventions: Behavioral: Postpartum Visit 3-4 Weeks
- Postpartum Visit 6-8 Weeks (Experimental): Participants will have postpartum visit scheduled 6-8 weeks after birth
  Interventions: Behavioral: Postpartum Visit 6-8 Weeks

INTERVENTIONS:
Behavioral: Postpartum Visit 3-4 Weeks — This visit will be the same as the standard of care postpartum visit, but it will be scheduled earlier.
  Arms: Postpartum Visit 3-4 Weeks
Behavioral: Postpartum Visit 6-8 Weeks — This standard of care postpartum visit will be scheduled for the standard time interval.
  Other Names: Standard of Care
  Arms: Postpartum Visit 6-8 Weeks

SUMMARY:
Due to potential to improve family planning, clinicians are increasingly interested in shortening the time to postpartum visits, but lack an evidence base to change policy.There are no studies that have examined the effectiveness of shortened interval to postpartum visit on attendance rate, contraception use, and rapid repeat of pregnancy (RROP). With this research, the investigators propose to conduct a randomized controlled trial (RCT) to examine the effect of reduced time interval to postpartum visit (3-4 weeks rather than 6-8 weeks) on postpartum visit attendance rate, contraceptive use, and RROP.

DETAILED DESCRIPTION:
Postpartum care is an essential component of women's reproductive health. During this time, the health care provider and the new mother review the previous pregnancy course, assess the mother's wellbeing, and establish treatment plans for any ongoing problems. Prospective guidance is given for both the mother and the baby in areas such as breastfeeding, nutrition, depression screening, and perineal/vulvar care. However, one of the most important goals of the postpartum visit is to discuss the new mother's desire for future pregnancies and the interval she wishes before another pregnancy. Inadequate reproductive health planning may result in unintended or rapid repeat of pregnancy (RROP), clinically defined as a second pregnancy within 24 months of the end of a previous pregnancy. A short inter-pregnancy interval is a risk factor for poor pregnancy outcomes including stillbirth, early neonatal death, extreme preterm births, and babies born small for gestational age. Compared to women who conceived 18-23 months after a previous birth, women conceiving less than five months after a previous birth had increased third trimester bleeding, uterine infection, premature rupture of membranes, and maternal death.Central to these outcomes is the rate of postpartum contraception use.

In fact, research shows an association between a postpartum visit and use of a reliable contraceptive method after pregnancy.

The optimal time for postpartum visit may be 3-4 weeks post-delivery rather than 6-8 weeks post-delivery with regard to visit attendance and proactive management of reproductive health, including contraception and time intervals between pregnancies. The timing of the postpartum visits are also linked to economic outcomes and healthcare utilization; postpartum care that results in decreased RROP and unintended pregnancies will likely decrease healthcare costs associated with the adverse consequences of inadequate reproductive health planning. Despite the obvious potential benefits of a decreased interval between delivery and the postpartum visit, to date, there have been no studies to systematically compare the impact of postpartum visit timing on visit attendance, contraception use and, subsequently, RROP.

This study is designed to investigate the effect of reduced time interval to postpartum visit on postpartum visit attendance rate, contraceptive use, and RROP. Additionally, the study will assess the impact of the two visit schedules on these outcomes by race, providing critical information about high risk populations. Finally, this research will assess the cost effectiveness of the shortened postpartum visit schedule relative to the standard of care. In order to account for potential bias in increased attendance rate due to intervention effect, compensation and other factors, this study will also compare the effectiveness of shortened time interval to postpartum visit on postpartum attendance rate and contraceptive use to a historic cohort.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* delivered vaginally a healthy, full-term (at least 37 weeks gestation) baby
* received prenatal care services at the VCUMCV OB clinic
* speak English
* provide informed consent for study participation.

Exclusion Criteria:

* cognitive impairment, psychiatric instability, or language barriers that limit their ability to provide informed consent
* surgically sterilized
* have complicated deliveries that require extended hospital stays
* need early follow-up to monitor their conditions
* any problems with infants such as preterm birth, admission to the Neonatal Intensive Care Unit (NICU), congenital malformations or respiratory problems that would require frequent clinic visits or prolonged hospital admissions for the infants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 364 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Postpartum Clinic Attendance | assessed at 12 weeks postpartum
  To compare the effectiveness of 3-4 week and 6-8 week intervals to postpartum visit on improving the rate of postpartum visit attendance. The investigators hypothesize that study participants with postpartum visits scheduled 3-4 weeks after delivery will be more likely to attend visits than study participants scheduled for visits 6-8 weeks after delivery.

SECONDARY OUTCOMES:
Contraception Use | Assessed at 3, 6, 9, 12, & 18 month follow-ups
  Compare the effectiveness of 3-4 week and 6-8 week intervals to postpartum visit on consistent contraceptive use
Rapid Repeat Pregnancy | Assessed at 3, 6, 9, 12, & 18 month follow-ups
  Compare the effectiveness of 3-4 week and 6-8 week intervals to postpartum visit on repeat pregnancy
Cost effectiveness | 18 month postpartum
  Compare overall cost of postpartum care

OTHER OUTCOMES:
Racial Differences | baseline, postpartum, 3, 6, 9, 12, & 18 month follow-ups
  Compare the effectiveness of 3-4 week and 6-8 week intervals to postpartum visit on reducing racial differences in postpartum visit attendance rates and contraceptive use. Specifically, the study team hypothesizes that the difference in postpartum visit attendance and consistent contraceptive use rates between AA and CA study participants will be lower among study participants with postpartum visits scheduled 3-4 weeks after delivery compared to study participants scheduled for visits 6-8 weeks after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Saba W Masho, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512
- [Derived] Masho SW, Ihongbe TO, Wan W, Graves WC, Karjane N, Dillon P, Bazzoli G, McGee E. Effectiveness of shortened time interval to postpartum visit in improving postpartum attendance: Design and rationale for a randomized controlled trial. Contemp Clin Trials. 2019 Jun;81:40-43. doi: 10.1016/j.cct.2019.04.012. Epub 2019 Apr 18. PMID 31004814